CLINICAL TRIAL: NCT02943668
Title: A Phase II Study of Deferasirox in Patients With Myelodysplastic Syndromes Who Are Anemic With Iron Overload
Brief Title: Deferasirox in Treating Patients With Very Low, Low, or Intermediate-Risk Red Blood Cell Transfusion Dependent Anemia or Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9422; NCI-2016-01457 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9422 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Results first posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-04

CONDITIONS: Anemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia; Myelodysplastic Syndromes | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (deferasirox) (Experimental): Patients receive deferasirox PO QD. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Deferasirox; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Deferasirox — Given PO
  Other Names: Exjade
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well deferasirox works in treating patients with very low, low, or intermediate-risk anemia or myelodysplastic syndrome that depends on red blood cell transfusions. Deferasirox may treat too much iron in the blood caused by blood transfusions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the activity of iron chelation therapy (ICT) with deferasirox, in patients with anemia due to myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

I. Reduction in red blood cell (RBC) transfusion requirements. II. Hematologic improvement. III. Change in serum ferritin levels from baseline to the end of the study as measured on a monthly basis.

IV. Safety and tolerability of deferasirox.

EXPLORATORY OBJECTIVES:

I. Blood and marrow samples will be taken to study erythropoiesis and the impact of iron overload on erythropoiesis.

OUTLINE: Patients receive deferasirox orally (PO) once daily (QD). Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving written informed consent prior to any study-specific procedures
* Diagnosis of MDS as defined by the World Health Organization (WHO) diagnostic criteria
* Have very low, low or intermediate-risk disease by the Revised International Prognostic Scoring System (IPSS-R)
* Baseline serum ferritin level >= 100 ng/mL
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Anemia defined as: hemoglobin =< 10.0 g/dL
* Bilirubin =< 1.5 times upper limit of normal (ULN)
* Alanine aminotransferase (ALT), and aspartate aminotransferase (AST) =< 3.5 times ULN
* Serum creatinine =< 1.5 x ULN
* Estimated glomerular filtration rate (GFR) > 40 mL/min
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the study and for 3 months following the last dose of deferasirox

  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using effective methods of contraception during dosing of study treatment; effective contraception methods include:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
    * Total abstinence or (when this is in line with the preferred and usual lifestyle of the subject); periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening); for female subjects on the study, the vasectomized male partner should be the sole partner for that subject
  * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential; sexually active males must use a condom during intercourse while taking drug and for 28 days after stopping study medication and should not father a child in this period; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
* Females with childbearing potential* must have had a negative urine or serum pregnancy test =< 7 days before the first dose of deferasirox and must also not be breastfeeding
* Reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* If the patient is currently receiving erythroid stimulating agents (ESA) with plans to continue during study, less than 2 months duration of ESA prior to starting study drug and no dose escalation within 2 months of start of study drug
* If the patient is being treated with granulocyte-colony stimulating factor (GCSF) and/or a TPO-mimetic (for example, eltrombopag or romiplostim) with plans to continue during the study: Less than 2 months duration of GCSF or the TPO-mimetic treatment prior to starting study drug; or GCSF and/or TPO-mimetic has been added to ESA therapy within 2 months of start of study drug
* If patient is being treated with lenalidomide with plans to continue during the study: Stable dose for less than 3 months prior to start of study drug
* If patient is being treated with hypomethylating agents (HMA) (for example, azacitidine or decitabine) with plans to continue during the study: Stable dose for less than 6 months prior to start of study drug
* Currently enrolled in, or discontinued within the last 14 days from a clinical trial involving an investigational product or non-approved use of a drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Presence of >= 10% blast by morphologic examination of bone marrow aspirate or biopsy
* Platelets =< 50,000
* Microcytosis on screening blood cell count (CBC) (mean corpuscular volume [MCV] < 81 fL)
* Active gastrointestinal (GI) ulceration or hemorrhage
* Have a serious preexisting medical condition that, in the opinion of the investigator would preclude participation in the study (for example a GI disorder causing clinically significant symptoms such as nausea, vomiting, and diarrhea, or malabsorption syndrome) or that would result in a life expectancy of less than 1 year
* Known hypersensitivity to deferasirox
* History of non-transfusional hemosiderosis
* Prior hematopoietic stem cell transplant for the diagnosis of MDS
* A second primary malignancy that in the judgment of the principal investigator (PI) or designee may affect the interpretation of results
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis
* Currently using aluminum-containing antacid products
* History of clinically significant auditory or ocular toxicity with ICT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Scott, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Deferasirox)
Started | 2
Completed | 1
Not Completed | 1
Not completed — Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Deferasirox)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients That Achieve Erythroid Hematologic Improvement.
Description: As defined by the modified International Working Group (IWG) response criteria:
  Erythroid response (pretreatment, <11 g/dL):
  1. Hgb increase by ≥ 1.5 g/dL
  2. Relevant reduction of units of RBC transfusions by an absolute number of at least 4 RBC transfusions/8 wk compared with the pretreatment transfusion number in the previous 8 wk. Only RBC transfusions given for a Hgb of ≤ 0.9 g/dL pretreatment will count in the RBC transfusion response evaluation.
  Platelet response (pretreatment, < 100 x 10^9/L)
  1. Absolute increase of ≥ 30 x 10^9/L for patients starting with > 20 x 10^9/L platelets
  2. Increase from < 20 x 10^9/L to > 20 x 10^9/L and by at least 100%
  Neutrophil response (pretreatment, < 1.0 x 10^9/L)
  1) At least 100% increase and an absolute increase > 0.5 x 10^9/L
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Deferasirox): Patients receive deferasirox PO QD. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Deferasirox: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Of the two participants on the study, none achieved erythroid hematologic improvement as defined by the modified IWG response criteria at 6 months.
Arm/Group | Treatment (Deferasirox)
Number analyzed (Participants) | 2
Participants | 0

2. Secondary Outcome: Change in Red Blood Cell (RBC) Transfusion Requirements
Description: Assessed monthly for up to twelve months.
Time Frame: Baseline up to 12 months
Population: Data for the 2 participants is presented as 2 different groups to show the individual RBC transfusion requirements per month, at each point in time
Measure: Number; unit: RBC transfusions/month
Groups:
- Patient 1; Patient 2: Patients receive deferasirox PO QD. Treatment continues for up to 52 weeks in the absence of disease progression or unacceptable toxicity.
  Deferasirox: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Patient 1 | Patient 2
Number analyzed (Participants) | 1 | 1
RBC transfusions/month
  Transfusion requirement at Baseline | 4 | 1
  Transfusion requirement at time off-treatment | 2 | 2

3. Secondary Outcome: Change in Serum Ferritin Levels
Description: Assessed monthly for up to twelve months.
Time Frame: Baseline up to 12 months
Population: Data for the 2 participants is presented as 2 different groups to show the individual serum ferritin levels at each point in time
Measure: Number; unit: ng/mL
Arm/Group | Patient 1 | Patient 2
Number analyzed (Participants) | 1 | 1
ng/mL
  Baseline | 6025 | 755
  1 month | 6637 | 778
  2 months | 6010 | 827
  3 months | 6405 | 583
  4 months | 22360 | 414
  5 months | 7252 | 652
  6 months | 5697 | 776
  7 months | 4832 | 880
  8 months | 4054 | NA — Patient went off-study after 7 months.
  9 months | 3933 | NA — Patient went off-study after 7 months.
  10 months | 3728 | NA — Patient went off-study after 7 months.
  11 months | NA — Patient went off-study after 10 months. | NA — Patient went off-study after 7 months.
  12 months | NA — Patient went off-study after 10 months. | NA — Patient went off-study after 7 months.

4. Secondary Outcome: Proportion of Patients Who Achieve Granulocyte or Platelet Hematologic Improvement
Description: as for outcome 1
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Deferasirox)
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: Enrollment through 30 days after the last administration of the study treatment
Arm/Group | Treatment (Deferasirox)
All-Cause Mortality (participants affected / at risk) | 1/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Deferasirox) (N=2)
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Deferasirox) (N=2)
Clostrid Difficile (Infections and infestations) | 1
Sinus Infection (Infections and infestations) | 1
Fracture- Lft. Lateral Tibia Plateau (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture- Lft. Second Metatarsal (Injury, poisoning and procedural complications) | 1
Fracture- Lft. Wrist (Injury, poisoning and procedural complications) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
A-fib w/ rapid ventricular rate (Cardiac disorders) | 1
Anemia- due to acute blood loss (Blood and lymphatic system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Weight loss (Investigations) | 1
Insomnia (Psychiatric disorders) | 1
Elevated Creatine/ urine protein (Renal and urinary disorders) | 1
Alanine Amniotransferase- increased (Investigations) | 1
Asparate Aminotransferase increased (Investigations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT02943668/Prot_SAP_000.pdf